CLINICAL TRIAL: NCT00621998
Title: A Randomized Controlled Trial of Risperidone and Olanzapine for the Schizophrenic Patients With Neuroleptic-Induced Tardive Dyskinesia
Brief Title: Risperidone and Olanzapine for the Schizophrenic Patients With Neuroleptic-Induced Tardive Dyskinesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan (Other Government)
Collaborators: Department of Health (Ambiguous)
Responsible Party: Hung-Yu Chan/ Attending Psychiatry and Director of General Psychiatry, Taoyuan Mental Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMH-91-02; DOH-890010
Record Dates: First submitted 2008-02-13; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2000-02

CONDITIONS: Neuroleptic-Induced Tardive Dyskinesia
Keywords: Risperidone; Olanzapine; Tardive dyskinesia
MeSH Terms: conditions — Tardive Dyskinesia | interventions — Risperidone; Olanzapine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Flexible dose of olanzapine
  Interventions: Drug: olanzapine
- 2 (Active Comparator): Flexible dose of risperidone
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: risperidone — 0.5-6 mg/day
  Arms: 2
Drug: olanzapine — 2.5-20 mg/day
  Arms: 1

SUMMARY:
We initiate a study with research grant from department of health and Taoyuan mental hospital and choose risperidone and olanzapine as study medications. We compare the effects of these 2 drugs in schizophrenic spectrum patients of Han ethnics with neuroleptic-induced tardive dyskinesia to test the hypothesis that these two medications have different effects in improving tardive dyskinesia.

DETAILED DESCRIPTION:
Objective: First generation antipsychotics would induce tardive dyskinesia in some schizophrenic patients. Second generation antipsychotics were the choices for these patients. But which one of second generation antipsychotic was the better choice did not have definitive results. We compared risperidone and olanzapine in schizophrenic patients with neuroleptic-induced tardive dyskinesia to see their effects in improving tardive dyskinesia. We also collected the data of average dose of risperidone and olanzapine to help the dosing strategy guidelines for the schizophrenic patients with neuroleptic-induced tardive dyskinesia.

Method: This randomized, rater-blind, parallel group, flexible dose study enrolled patients from Taoyuan Mental Hospital from July 2000 to December 2003. Schizophrenia, schizophreniform or schizoaffective disorder (DSM-IV) patients who met the research criteria of neuroleptic-induced tardive dyskinesia research criteria of DSM-IV and no less than moderate severity (> or =4) of global impression of extrapyramidal syndrome rating scale (ESRS). 60 patients were random assignment to risperidone or olanzapine for 24 weeks. The primary outcome was to compare the change of total scores of abnormal involuntary movement scale from baseline to study endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18-70 y/o
* Female patients did not have pregnancy plans and must agree to use reliable pregnancy prevention methods if during childbearing age
* Meet schizophrenia, schizophreniform or schizoaffective disorder criteria of DSM-IV
* Fulfill DSM-IV neuroleptic-induced tardive dyskinesia research criteria, the severity of tardive dyskinesia was no less than moderate degree (> or =4) assessed by global impression of Extrapyramidal System Rating Scale (item 42 of ESRS)
* Patients or legal responsible people agree to join study and sign informed consent

Exclusion Criteria:

* Had other axis I diagnosis of DSM-IV
* Unstable major systemic diseases
* Had neurological disorder influenced to EPS assessment
* Substance abuse or dependence other then coffee or tobacco within 6 months before study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2000-07; Primary Completion 2003-12 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Total scores of AIMS | The change from baseline to study endpoint

SECONDARY OUTCOMES:
Total scores of BPRS | The change from baseline to study endpoint
Extrapyramidal syndrome rating scale | The change from baseline to study endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Yu Chan, M.D., M.S., Study Chair — Taoyuan Psychiatric Center, Ministry of Health and Welfare, Executive Yuan, R.O.C. Taiwan
Locations (1):
- Taoyuan Mental Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chan HY, Chiang SC, Chang CJ, Gau SS, Chen JJ, Chen CH, Hwu HG, Lai MS. A randomized controlled trial of risperidone and olanzapine for schizophrenic patients with neuroleptic-induced tardive dyskinesia. J Clin Psychiatry. 2010 Sep;71(9):1226-33. doi: 10.4088/jcp.09m05155yel. PMID 20441726